CLINICAL TRIAL: NCT06265545
Title: Multicenter, Platform-type Clinical Study of Refractory/Recurrent Acute Myeloid Leukemia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: IIT2024001
Record Dates: First submitted 2024-01-17; First posted 2024-02-20 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: AML; Refractory; Relapsed
Keywords: AML; Refractory; Relapsed
MeSH Terms: conditions — Recurrence | interventions — ivosidenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- Arm 1 (Experimental): With IDH1 gene mutation(up to 2 cycles available):IVA :
  Ivosidenib 500mg d1-28 Azacitidine 75mg/m2/d d1-7 Venetoclax100mg d1,200mg d2,400mg d3-21 400mg ;d22-28(If the proportion of 21st bone marrow blasts is greater than 5%)
  Interventions: Drug: Ivosidenib,Venetoclax,gilteritinib,Selinexor
- Arm 2 (Experimental): FLT3/ITD or FLT3/TKD gene mutation (up to 2 cycles available)
  GV :
  Gilteritinib 120mg, d1-28 Venetoclax 100mg d1, 200mg d2, 400mg d3-21 400mg d22-28 (if the proportion of 21st bone marrow blasts are greater than 5%)
  Interventions: Drug: Ivosidenib,Venetoclax,gilteritinib,Selinexor
- Arm 3 (Experimental): For R/R AML patients without IDH1 or FLT3 mutations who have not been exposed to Venecra in the last 3 months, the investigators will determine whether they are fit patients based on physical status and comorbidivities, and if they are, they can be randomly assigned to Arm3 or Arm4 DAV/IAV/MAV Cytarabine 100mg/m2/d, d1-5 Daunorubicin 60mg/m2/d, d1-2, or Idarubicin 12mg/m2/d, d1-2, or mitoxantrone 8mg/m2/d d1-2 Venetoclax 100mg d3, 200mg d4, 400mg d5-11;
  Interventions: Drug: Ivosidenib,Venetoclax,gilteritinib,Selinexor
- Arm 4 (Experimental): HAV :
  Cytarabine 100mg/m2/d, d1-5 Homoharringtonine 2mg/m2 d1-5 Venetoclax 100mg d3, 200mg d4, 400mg d5-11
  Interventions: Drug: Ivosidenib,Venetoclax,gilteritinib,Selinexor
- Arm 5 (Experimental): A patient with R/R AML without IDH1 or FLT3 mutation who has not been exposed to Venetoclax in the last 3 months but who is judged by the investigators to be unfit based on physical fitness and comorbidivities is unfit to enter Arm5.
  Arm5: (up to 4 cycles available)
  VA :
  Azacytidine 75mg/m2/d d1-7 Venetoclax 100mg d1, 200mg d2, 400mg d3-21 400mg d22-28 (if the proportion of 21st bone marrow blasts are greater than 5%)
  Interventions: Drug: Ivosidenib,Venetoclax,gilteritinib,Selinexor
- Arm 6 (Experimental): Patients with R/R AML without IDH1 or FLT3 mutations who have been exposed to Vinecra within the last 3 months may be enrolled in the exploratory protocol group based on a comprehensive assessment of local drug availability and patient status:
  Arm6:
  The Investigator's choice (IC) option involves a range of drugs such as clatabine, PI3K inhibitors, histone deacetylase inhibitors, celinisol, and novel liposomes.
  Interventions: Drug: Ivosidenib,Venetoclax,gilteritinib,Selinexor
- Arm 7 (Experimental): According to the patient's condition and physical condition, evaluate whether there is a suitable new drug clinical trial to be enrolled. If there is, enter the Arm 7 (new drug clinical trial).
  Interventions: Drug: Ivosidenib,Venetoclax,gilteritinib,Selinexor

INTERVENTIONS:
Drug: Ivosidenib,Venetoclax,gilteritinib,Selinexor — if the target gene mutations are positive, enter arm1 or arm2. other conditions, enter the chemotherapy arms (Arm3-6)

SUMMARY:
To study the optimal therapeutic strategies for salvage treatment of refractory/relapsed AML, and to clarify the effectiveness and safety of various salvage treatment options. A prospective, multicenter, platform-type study was conducted to explore the overall response rate, tolerability, and survival of patients with R/R AML with different treatment regimens.

DETAILED DESCRIPTION:
It is recommended to routinely screen for chromosomal karyotype, FLT3/ITD, FLT3/TKD and IDH1 mutations before enrollment.According to the patient's condition and physical condition, evaluate whether there is a suitable new drug clinical trial to enroll, if there is, enter the Arm 7 (new drug clinical trial); If not, enter other arm of the clinical study.According to the results of gene mutation, patients with target gene mutations should enter the corresponding study cohort (Arm1, Arm2), and select the regimen of specific targeted drug composition. For patients without a target mutation, patients eligible for intensive chemotherapy who had not received Venetoclax in the last 3 months were randomized to the Daunorubicin/idarbicin/mitoxantrone combination cytarabine + Venetoclax(DAV) (Arm3) and the Hyperhardinine combination cytarabine + Venetoclax cohort (HAV) (Arm4). Patients who were intolerant to intense chemotherapy were enrolled in the Venetoclax combined with Azacitidine cohort (Arm5). For patients who have failed treatment with Venetoclax within the last 3 months, the Venetoclax-based regimen is not recommended again and the physician is advised to conduct an exploratory trial (Arm6). After CR form induction therapy, allogeneic hematopoietic stem cell transplantation should be selected as far as possible according to the patient's wishes. For patients who are unable or unwilling to undergo allogeneic hematopoietic stem cell transplantation, physicians may choose post-remission consolidation therapy based on experience.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients with acute myeloid leukemia (except for acute promyelocytic leukemia) diagnosed by bone marrow cell morphology, immunology and genetics above are classified according to the French-British-American Collaboration diagnostic criteria (FAB criteria) and the World Health Organization diagnostic criteria (WHO2016 criteria).

  2. Meet criteria for refractory/recurrent AML (except APL). The recurrence was morphological recurrence, excluding molecular recurrence. Except for simple extramedullary leukemia.

  3. Age and gender are not limited. 4. Informed consent must be signed before the start of the study procedure, and the informed consent must be signed by the patient himself or his immediate family if he is 18 years old and above; For young patients under the age of 18, the legal guardian shall sign the informed consent. Considering the patient's condition, if the patient's signature is not conducive to the treatment of the condition, the informed consent shall be signed by the legal guardian or the patient's immediate family.

Exclusion Criteria:

1. Concurrent malignant tumors of other organs (patients requiring treatment).
2. Participants considered unsuitable for inclusion by the researchers.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-02-22 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Complex response (CRc) rate (including CR and CRi) | Time from remission date of the first subject until remission date of the last subject.
  Proportion of patients with combined responses (complete and partial responses)

SECONDARY OUTCOMES:
mortality associated with salvage treatment (30 days, 60 days) | Treatment within 30 days and 60 days
  Mortality of patients treated within 30 and 60 days
MRD-negative complete response rate | the whole period of the trial, up to 730 days
  Proportion of patients with complete response and MRD negative
Overall survival | the whole period of the trial, up to 730 days
  Used to evaluate all patients entering clinical trials
Event-free survival | the whole period of the trial, up to 730 days
  It is only used to evaluate patients who have achieved CR
Relapse-free survival | the whole period of the trial, up to 730 days.
  It is only used to evaluate patients who have achieved CR

CONTACTS AND LOCATIONS:
Locations (1):
- Blood Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No